CLINICAL TRIAL: NCT07091110
Title: Efficacy of LigaSure Versus Harmonic Scalpel US in Laparoscopic Appendectomy in Management of Acute Appendicitis
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed I Farid, assistant professor of general surgery, Zagazig University
Other Study IDs: ZU-IRB#1419/17-6-2025
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Appendicitis Acute
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- A: laparoscopic appendectomy using harmonic US scalpel and endoloop
  Interventions: Procedure: laparoscopic appendectomy
- B: Laparoscopic appendectomy using LigaSure plus endoloop
  Interventions: Procedure: laparoscopic appendectomy

INTERVENTIONS:
Procedure: laparoscopic appendectomy — laparoscopic appendectomy

SUMMARY:
Background Acute appendicitis is the most frequent abdominal surgical emergency worldwide, peaking in incidence between the second and third decade of life. Appendectomy was the only treatment for appendicitis for more than a century, and it is still the most common treatment. The surgical treatment for appendicitis is an appendectomy, which can be performed laparoscopically or openly. The purpose of the current study is to determine and measure the safety and effectiveness of laparoscopic appendectomy with LigaSure and harmonic US scalpels.

Patients and methods:

This research was carried out from January 2023 to January 2025, involved 60 patients who complained of acute lower abdominal pain in their right side, and were diagnosed with suspected acute appendicitis. Two groups of patients were formed: Group A had an appendectomy performed laparoscopically using a harmonic US scalpel, and group B underwent a laparoscopic appendectomy using LigaSure.

DETAILED DESCRIPTION:
Study Design This is a prospective comparative study for a total of 60 patients participated in this study, which ran from January 2023 to January 2025. Patients were complaining of acute right lower abdominal pain, after clinical examination, laboratory and radiological investigations diagnosed as acute appendicitis. Patients were randomized by the closed envelope method into 2 equal groups; 30 patients for each. Group A (laparoscopic appendectomy using harmonic US scalpel and endoloop) and group B (laparoscopic appendectomy using LigaSure plus endoloop).

Study Approval Ethical approval for this study was granted by the Institutional Review Board of the Zagazig University, with an IRB registration number is ZU-IRB#1419/17-6-2025.

Inclusions criteria This study included 26 female and 34 male patients. All patients presented with clinically, laboratory and radiographically confirmed acute appendicitis. All of whom were between the ages of 18 and 60.

Exclusions criteria We excluded patients with complicated acute appendicitis as appendicular mass or abscess, patients with history of previous multiple open abdominal surgeries, patients with economic factors and also patients who preferred conventional, open appendectomy to laparoscopic removal approach.

Examination, diagnosis and Workup protocol The patient's complete medical history (including a typical recent non-neglected right lower abdomen or periumbilical discomfort, nausea/vomiting, anorexia, or a low grade fever, etc.) and physical examination (right iliac fossa tenderness or guarding with a positive Mc-Burney's sign, cough test, etc.) were used to make the clinical diagnosis of non-complicated acute appendicitis. Laboratory tests such as the complete blood count (CBC), C-reactive protein (CRP), pregnancy test for female patients in the childbearing age range, etc., were needed for each patient and interpreted. Additionally, all patients underwent an ultrasound, either with or without a pelvi-abdomen CT scan with contrast, to confirm the diagnosis, rule out other potential causes of acute abdomen, and-most importantly-rule out patients with complicated appendicitis, such as those with phlegmon, generalized peritonitis, or appendicular abscess.

Following an explanation on the diagnosis, the steps involved in the laparoscopic procedure, the benefits, dangers, and potential issues, all patients who satisfied the criteria for surgery were given written consent. The patient was placed on IV fluids, prophylactic broad-spectrum IV antibiotics (Ceftriaxone 2g IV), and NPO as part of the operation, which was completed within 24 hours of the diagnosis and management.

The Surgical Procedure The procedure was carried out with the patient in a supine position under general anesthesia. After the abdomen was prepared and wrapped, three trocars were placed inside of it. Using a laparoscopic Veress needle, the first trocar (10mm) for pneumoperitoneum (figure 1) was inserted in the periumbilical region. In the right or the left iliac fossa (according to the intraoperative position of the appendix and the surgeon preference), is the second trocar 5 mm functioning port. Third trocar 5 mm functioning port located above the pubic area (figure 2).

Diagnose the appendix, examine for any pathology, and then begin the procedure. Ligation of the base using endoloops(figure 3), coagulation, sealing, and division of the mesoappendix using either ligaSure (figure 4) or Harmonic US (figure 5) as the energy source. Under direct vision, all of the trocars were extracted while the abdomen was deflated. Layers of skin closure using Monocryl 4/0 for both modules of the procedure. Following surgery, all specimens were sent for histological analysis.

The operating nurse noted the duration of each group's operation. Twelve hours after surgery, all patients were put on a liquid diet and given little sips of water. Only in cases where the appendix was significantly inflamed or perforated were antibiotics administered for at least three days after surgery. Early ambulation was advised for all patients in order to assist bowel movements. Both groups of patients were released from the hospital 1 to 2 days following surgery.

Statistical analysis The categorical variables were presented as a number (%), while the continuous variables were presented as the mean ± SD & median (range). Using the Shapiro-Wilk test, continuous variables were examined for normality. Separate samples two groups of regularly distributed data were compared using the Student's t-test, and non-normally distributed variables were compared using the Mann Whitney U test. When appropriate, Fisher's exact test or Pearson's chi-square test were used to compare the percentage of categorical variables. Every test had two tails. It was deemed statistically significant when the P-value was less than 0.05. SPSS version 22.0 for Windows (IBM Corp., Armonk, NY, USA) was used for all statistics

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria This study included 26 female and 34 male patients. All patients presented with clinically, laboratory, and radiographically confirmed acute appendicitis. All of whom were between the ages of 18 and 60.

Exclusion Criteria:

* We excluded patients with complicated acute appendicitis, such as appendicular mass or abscess, patients with a history of previous multiple open abdominal surgeries, patients with economic factors, and also patients who preferred conventional, open appendectomy to the laparoscopic removal approach.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This is a prospective comparative study for a total of 60 patients participated in this study, which ran from January 2023 to January 2025. Patients were complaining of acute right lower abdominal pain, after clinical examination, laboratory and radiological investigations diagnosed as acute appendicitis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
the average range of operating time for both groups | from January 2023 to January 2025
  Depending on the degree of difficulties experienced, the average range of operating time for both groups was reported.

SECONDARY OUTCOMES:
intraoperative complications | from January 2023 to January 2025
  In both groups, any intraoperative complications, such as haemorrhage, bowel or organ damage is recorded
conversion to open surgery | from January 2023 to January 2025
  any case is discovered to have difficult appendicitis during surgery, either with early appendicular phlegmon or with an appendicular abscess with minor collections, conversion to open surgery is documented.
postoperative complications | from January 2023 to January 2025
  any case with postoperative complications, as bleeding, infection, or collection is reported

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided